CLINICAL TRIAL: NCT00485693
Title: A Phase 2 Multicenter, Randomized, Double-blind, Parallel-group, Active-control, Dose-ranging Study to Evaluate the Safety, Efficacy, and Comparative Systemic Bioavailability of a Single Administration of SKY0402 Via Local Infiltration for Prolonged Postoperative Analgesia in Subjects Undergoing Total Knee Arthroplasty.
Brief Title: Dose-Ranging Study for Prolonged Postoperative Analgesia in Subject Undergoing Total Knee Arthroplasty
Acronym: TKA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SKY0402C208
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Postoperative Pain
Keywords: pain; postoperative; total knee arthroplasty; analgesia
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine HCl (Active Comparator): Bupivacaine HCl (Marcaine 0.25% with epinephrine 1:200,000)
  Interventions: Drug: Bupivacaine HCl
- SKY0402 (Other): SKY0402 at various dosage levels. Single administration.
  Interventions: Drug: SKY0402

INTERVENTIONS:
Drug: Bupivacaine HCl — 150 mg Bupivacaine HCl
  Other Names: Bupivacaine HCl (Marcaine 0.25% with epinephrine 1:200,000)
  Arms: Bupivacaine HCl
Drug: SKY0402 — 600 mg SKY0402 (study drug)
  Other Names: EXPAREL
  Arms: SKY0402

SUMMARY:
Dose-ranging study for prolonged postoperative analgesia in subjects undergoing total knee arthroplasty

DETAILED DESCRIPTION:
This is a phase 2, multicenter, parallel-group, active-control, randomized, double-blind, dose-ranging study conducted to evaluate three dose levels of SKY0402 compared with 150 mg of bupivacaine HCl.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, greater than or equal to 18 and less than or equal to 75 years of age at the Screening Visit.
2. Female subjects only: Postmenopausal, surgically sterile, or willing to use acceptable means of contraception for at least 30 days after surgery including any of the following: hormonal contraceptives (e.g., oral, injectable, implantable starting at least 30 days before study drug administration), effective double-barrier methods (e.g., condoms with spermicide), intrauterine device, lifestyle with a personal choice of abstinence, nonheterosexual lifestyle, or a strictly monogamous relationship with a partner who has had a vasectomy.
3. Scheduled to undergo primary unilateral total knee arthroplasty (TKA) under general anesthesia.
4. American Society of Anesthesiology (ASA) Physical Class 1-3.
5. Able and willing to comply with all study visits and procedures.
6. Able to speak, read, and understand the language of the Informed Consent, study questionnaires, and other instruments used for collecting subject-reported outcomes, in order to enable accurate and appropriate responses to pain scales and other required study assessments.
7. Willing and capable of providing written informed consent.

Exclusion Criteria:

1. Pregnancy, nursing, or planning to become pregnant during the study or within one month after dosing.
2. Use of any of the following medications within the times specified before surgery:

   * Long-acting opioid medication within 3 days.
   * Any opioid medication within 24 hours.
3. Concurrent, painful, physical condition or concurrent surgery that may require analgesic treatment in the postoperative period for pain that is not strictly related to the surgical site administered study treatment, and which may confound the postoperative assessments (e.g., significant pain from other joints, chronic neuropathic pain, concurrent contralateral TKA, concurrent foot surgery, etc.).
4. Body weight less than 50 kilograms (110 pounds) or morbid obesity.
5. Contraindication to any of the pain-control agents planned for postoperative use (e.g., acetaminophen, morphine, oxycodone, ketorolac).
6. Contraindication to epinephrine, such as concurrent administration of monoamine oxidase (MAO) inhibitors or antidepressants of amitriptyline or imipramine types, conditions where the production or exacerbation of tachycardia could prove fatal (e.g., poorly controlled thyrotoxicosis or severe heart disease), or any other pathological conditions that might be aggravated by the effects of epinephrine.
7. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.
8. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
9. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, may interfere with study assessments or compliance.
10. Current or historical evidence of any clinically significant disease or condition, especially cardiovascular or neurological conditions that, in the opinion of the Investigator, may increase the risk of surgery or complicate the subject's postoperative course.
11. Significant medical conditions or laboratory results that, in the opinion of the Investigator, indicate an increased vulnerability to study drugs and procedures, and expose the subject to an unreasonable risk as a result of participating in this clinical trial, such as: debilitating diseases, acute illnesses, hypotension, partial or complete conduction block, impaired cardiac function, untreated hypertension, advanced arteriosclerotic heart disease, cerebral vascular insufficiency, pre-existing abnormal neurological or neuromuscular disease (e.g., epilepsy, myasthenia gravis), advanced liver disease, severe renal impairment, advanced diabetes comorbid conditions associated with an immunocompromised status, such as blood dyscrasias, HIV/AIDS, or recent chemotherapy.

    In addition, the subject will be ineligible to receive study drug if he or she meets the following criteria during surgery:
12. Any clinically significant event or condition uncovered during surgery(e.g., excessive bleeding), which occurs before study drug administration, that might render the subject medically unstable or complicate the subject's postoperative course.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2007-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Davis, RN, Study Director — Pacira Pharmaceuticals, Inc
Locations (9):
- United States (6):
  - West Alabama Research, Inc., Birmingham, Alabama
  - California Clinical Research, Inc., Davis, California
  - Accurate Clinical Trials, Inc., Laguna Hills, California
  - St. Luke's Roosevelt Hospital, New York, New York
  - The Ohio State University Medical Center, Columbus, Ohio
  - Texas Tech University Health Science Center, Lubbock, Texas
- Czechia (3):
  - Urazova Nemocnice Brno, Brno
  - Regional Hospital Kladno, Kladno
  - The Hospital Trebic, Třebíč

REFERENCES:
- [Derived] Dasta J, Ramamoorthy S, Patou G, Sinatra R. Bupivacaine liposome injectable suspension compared with bupivacaine HCl for the reduction of opioid burden in the postsurgical setting. Curr Med Res Opin. 2012 Oct;28(10):1609-15. doi: 10.1185/03007995.2012.721760. Epub 2012 Sep 3. PMID 22900785

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine HCl; SKY0402: A single dose of study drug was to be administered intraoperatively via local infiltration
Period: Overall Study
Arm/Group | Bupivacaine HCl | SKY0402
Started | 34 | 104
Completed | 34 | 104
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine HCl | SKY0402 | Total
Number analyzed (Participants) | 34 | 104 | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 67 | 89
  >=65 years | 12 | 37 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (7.2) | 62.3 (7.4) | 62.2 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 62 | 85
  Male | 11 | 42 | 53
Region of Enrollment [Number; unit: participants]
  United States | 28 | 69 | 97
  Czech Republic | 6 | 35 | 41

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) With Activity (NRS-A) Pain Intensity Scores Through Postoperative Day 4
Description: The subject's pain intensity was to be assessed with activity (NRS-A) after actively flexing the involved knee to the maximum flexion point possible. The subject was asked to respond to the following question: "On a scale of 0 to 10, where 0 = no pain and 10 = worst possible pain, how much pain did you have while bending your knee?"
Time Frame: 0 to 96 hours
Measure: Mean (Standard Deviation); unit: Units on a scale*hours
Groups:
- Bupivacaine HCl: Single administration of 150 mg bupivacaine HCl in a 60-mL injection volume (undiluted)
- SKY0402 Low Dose: Single administration of SKY0402150 mg in a volume of 60 mL via local infiltration
- SKY0402 Low-mid Dose: Single administration of SKY0402 300mg in a volume of 60 mL via local infiltration
- SKY0402 High-mid Dose: Single administration of SKY0402 450 mg in a volume of 60 mL via local infiltration
- SKY0402 High Dose: Single administration of SKY0402 600mg in a volume of 60 mL via local infiltration
Arm/Group | Bupivacaine HCl | SKY0402 Low Dose | SKY0402 Low-mid Dose | SKY0402 High-mid Dose | SKY0402 High Dose
Number analyzed (Participants) | 34 | 28 | 25 | 26 | 25
Units on a scale*hours | 20.4 (3.9) | 20.7 (5.4) | 19.5 (5.3) | 18.8 (5.3) | 19.1 (4.4)

2. Secondary Outcome: Number of Participants With Adverse Events or Serious Adverse Events Through 30 Days
Time Frame: Up to 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Bupivacaine HCl | SKY0402
All-Cause Mortality (participants affected / at risk) | 1/34 | 1/104
Serious Adverse Events (participants affected / at risk) | 3/34 | 5/104
Other Adverse Events (participants affected / at risk) | 29/34 | 83/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine HCl (N=34) | SKY0402 (N=104)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine HCl (N=34) | SKY0402 (N=104)
Nausea (Gastrointestinal disorders) | 23 | 48
Constipation (Gastrointestinal disorders) | 13 | 36
Vomiting (Gastrointestinal disorders) | 6 | 16
Pyrexia (General disorders) | 11 | 38
Oedema peripheral (General disorders) | 11 | 30
Fatigue (General disorders) | 4 | 5
Hypotension (Vascular disorders) | 12 | 21
Dizziness (Nervous system disorders) | 6 | 13
Somnolence (Nervous system disorders) | 1 (1) | 11
Headache (Nervous system disorders) | 2 | 5
Lethargy (Nervous system disorders) | 0 (0) | 7
Anaemia postoperative (Injury, poisoning and procedural complications) | 7 | 13
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 8 | 25
Anaemia (Blood and lymphatic system disorders) | 6 | 16
Tachycardia (Cardiac disorders) | 4 | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 6
Pruritis (Skin and subcutaneous tissue disorders) | 6 | 10
Insomnia (Psychiatric disorders) | 5 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No